CLINICAL TRIAL: NCT01809340
Title: An Exploratory, Blinded, Randomized, Placebo-controlled Study in Subjects With Depressive Disorder to Investigate the Effect of Minocycline on Relapse After Successful Intravenous Ketamine/Minocycline-induced (Partial) Symptoms Response
Brief Title: The Effect of Minocycline on Relapse After Successful Intravenous Ketamine/Minocycline-induced Symptoms Response in Subjects With Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study team decision because of IP supply issue and necessary amendment to protocol
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100957; KETIVEDI2001 (Other: Janssen Research & Development, LLC); 2012-002954-21 (EudraCT Number)
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Depressive Disorder
Keywords: Depressive Disorder; Major Depressive Disorder; Depression; Bipolar Disorder Type II; Anti-depressant; Ketamine; Minocycline
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Depression; cyclopia sequence | interventions — Minocycline; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Minocycline (Experimental): Following a 12-day open-label treatment phase (involving ketamine and minocycline), responders may receive oral minocycline twice daily for up to 6 weeks in a blinded manner. In addition, non-responders may receive oral minocycline twice daily for up to 6 weeks in an open-label manner.
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator): Following a 12-day open-label treatment phase (involving ketamine and minocycline), responders may receive placebo twice daily for up to 6 weeks in a blinded manner
  Interventions: Drug: Placebo
- Ketamine and Minocycline (Experimental): All patients will receive 6 IV infusions of ketamine and oral minocycline twice daily during a 12-day open-label treatment phase
  Interventions: Drug: Minocycline; Drug: Ketamine

INTERVENTIONS:
Drug: Minocycline — In the 12-day open-label treatment phase, patients will self administer oral minocycline 200 mg on Day 1, 100 mg twice daily on Days 2 to 11, and 100 mg on the morning of Day 12. In the 6-week blinded treatment phase, responders may self administer oral minocycline 100 mg twice daily from the evening of Day 12 for up to 6 weeks (Day 54), or until relapse, whichever comes first. In the 6-week open-label treatment phase, non-responders may self administer oral minocycline 100 mg twice daily from the evening of Day 12 for up to 6 weeks (Day 54).
  Arms: Ketamine and Minocycline; Minocycline
Drug: Placebo — Patients in the 6-week blinded treatment phase, may self administer placebo twice daily from the evening of Day 12 for up to 6 weeks (Day 54), or until relapse, whichever comes first.
  Arms: Placebo
Drug: Ketamine — In the 12-day open-label treatment phase, all patients will receive 1 IV infusion of 0.5 mg/kg ketamine over 40 minutes on Days 1, 3, 5, 8, 10 and 12.
  Arms: Ketamine and Minocycline

SUMMARY:
The purpose of this study is to assess whether the antidepressant effect from intravenous (IV) ketamine treatment can be maintained by minocycline compared to placebo after IV ketamine treatment is stopped.

DETAILED DESCRIPTION:
This is a placebo-controlled (i.e., an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), double-blind (neither physician nor patient knows the treatment that the patient receives) randomized (the drug is assigned by chance) study in patients with Major Depressive Disorder (MDD) and Bipolar Disorder Type II. The study is designed to assess whether the antidepressant response to treatment with intravenous (IV) ketamine can be maintained by treatment with minocycline in patients with MDD and Bipolar Depression Type II (compared to placebo). Both hospitalized patients as well as patients being treated as an outpatient for their current episode of depression can qualify for participation in this study. The study has four sequential phases: if eligibility for the study has been confirmed during the 21-day screening phase, the patients will enter a 12-day open-label (ie, patient and physician know the intervention that is being administered) treatment phase during which the patient will receive 6 open-label IV infusions of 0.5 mg/kg ketamine on Day 1, 3, 5, 8, 10 and 12 in combination with open-label minocycline, orally administered twice daily. All patients will remain at the study site for at least 4 hours after the IV ketamine administrations. Response to treatment will be assessed using the Montgomery-Asberg Depression Rating Scale (MADRS) which is designed to measure the overall severity of depressive symptoms. Patients responding to ketamine/minocycline treatment will be randomized to receive minocycline or placebo for 6 weeks during a 6-week blinded treatment phase or until relapse. A patient will be defined as a "ketamine responder" if there is a 50% or more decrease in comparison to baseline values (Day 1 predose) in the MADRS total score performed at 3 to 4 hours postdose on Days 8, 10, or 12, with a 40% or more decrease from baseline in the MADRS total score on Day 12. Patients not responding to treatment with ketamine/minocycline will be given the option to receive 100 mg minocycline twice daily as open-label treatment for a maximum of 6 weeks. The patients (both responders and non-responders) will have weekly visits following last dose of ketamine until Day 54 (responders/non-responders) or until relapse (responders) whichever comes first, to determine the duration of the antidepressant effect and to assess safety and tolerability after completion of treatment. Upon completion of the study (Day 54) or at time of relapse all patients will have an end-of-study visit. All patients can return to standard of care treatment at the end of the study. The total study duration for each patient will be maximally 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria for moderate to severe major depressive disorder (MDD), without psychotic features, or Bipolar Disorder Type II
* Patients should have an Inventory of Depressive Symptomatology-Clinician Rated (IDS-C30) total score ≥ 34 at Screening and at Day 1 (predose)
* Patients with major depressive disorder should have failed at least two adequate treatment courses (dose and duration) with antidepressant therapy, one of which is in the current episode
* Patients should not have received electroconvulsive therapy (ECT) in the current episode but could be those for whom ECT is considered
* Patients with bipolar depression (BPD) Type II must have been taking a stable dose of a mood-stabilizing medication (e.g., lithium, valproate, carbamazepine, lamotrigine, antipsychotic agents) for at least 4 weeks, dosed clinically to target the therapeutic range
* Patients currently taking an antidepressant(s) must have received at least 2 weeks of stable antidepressant therapy at the time of Screening
* Doses of current antidepressant therapies should remain the same for the duration of the study
* Women must be postmenopausal, surgically sterile, or if heterosexually active, practicing a highly effective method of birth control
* Men who are heterosexually active with a woman of childbearing potential must agree to use a double barrier method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Has a current DSM-IV axis I diagnosis other than MDD or BPD Type II at screening (except for co-morbid anxiety disorders)
* Has a diagnosis of substance abuse or dependence within 6 months prior to screening evaluation (nicotine and caffeine dependence are not exclusionary)
* Patient is currently taking more than 4 psychotropic medications at Day 1 (predose)
* Has an autoimmune disorder such as Crohn's disease, rheumatoid arthritis, psoriasis currently treated with/requiring treatment with immunomodulatory therapies
* Has any significant cardiovascular, respiratory, neurologic, renal, hepatic, endocrine, or immunologic diseases based on screening examination
* Has uncontrolled hypertension (diastolic blood pressure ≥ 90 mmHg), despite diet, exercise or a stable dose of an allowed antihypertensive treatment, at Screening or Day 1 (predose)
* Has planned vaccination within 2 weeks prior to the first dose of study medication through 2 weeks after the last dose of study medication - Has an active infectious disease/current infection
* Has known allergies, hypersensitivity, or intolerance to minocycline or ketamine or its excipients - Has contraindications to the use of minocycline or ketamine per local prescribing information

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients (among responders) who survive relapse-free | Day 54
  The Montgomery-Asberg Depression Rating Scale (MADRS) measures depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition. Relapse is defined as MADRS ≥ 30.

SECONDARY OUTCOMES:
Change in MADRS total score among non-responders from pre-randomization to end-of-study | From Day 12 to Day 54
  The Montgomery-Asberg Depression Rating Scale (MADRS) measures depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Change in the MADRS total score from baseline during IV ketamine treatment phase | Days 1, 3, 5, 8, 10 and 12
  The Montgomery-Asberg Depression Rating Scale (MADRS) measures depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Change in the MADRS total score from baseline after IV ketamine treatment phase | Days 1, 20, 27, 34, 41, 48, and 54
  The Montgomery-Asberg Depression Rating Scale (MADRS) measures depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Response (reduction ≥ 50% in MADRS total score relative to baseline) rate during IV ketamine treatment phase | Days 1, 3, 5, 8, 10, and 12
  The Montgomery-Asberg Depression Rating Scale (MADRS) measures depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Time to relapse (among responders) following completion of the IV ketamine infusion schedule and after first dose of minocycline/placebo | From Day 12 to Day 54
  The Montgomery-Asberg Depression Rating Scale (MADRS) measures depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition. Relapse is defined as MADRS ≥ 30.
Change in C-SSRS from baseline to any time in the study | Days 1, 12, and 54
  The Columbia Suicide Severity Rating Scale (C-SSRS) is a clinical interview to assess severity and track suicidal events providing a summary of both suicidal ideation and behavior to identify the level and type of suicidality present.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (12):
- Belgium (3):
  - Duffel
  - Lede
  - Leuven
- France (3):
  - Besançon
  - Clermont-Ferrand
  - Nîmes
- Leiden, Netherlands
- Spain (5):
  - Alicante
  - Barcelona
  - Coslada
  - Madrid
  - Zamora

REFERENCES:
- See also: An exploratory, blinded, randomized, placebo-controlled study in subjects with depressive disorder to investigate the effect of minocycline on relapse after successful intravenous ketamine/minocycline-induced (partial) symptoms response — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3625&filename=CR100957_CSR.pdf